CLINICAL TRIAL: NCT06671977
Title: Phase 1 Study of the Safety, Tolerability, Electrophysiological Effects and Efficacy of DMT in Humans
Brief Title: Study of the Safety, Tolerability, Electrophysiological Effects and Efficacy of DMT in Humans
Acronym: DMT-Bolus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Deepak C. D'Souza (Other)
Responsible Party: Sponsor-Investigator, Deepak C. D'Souza, Deepak Cyril D'Souza, MD, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000034770
Record Dates: First submitted 2024-10-16; First posted 2024-11-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Major Depression Disorder; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Healthy individuals and individuals with current major depression will participate in 2 dosing sessions separated by 4 weeks, during which they will receive placebo, low dose DMT, medium dose DMT, low dose THC and medium dose THC. Subjects will be prepared for the dosing session and also debriefed after each dosing session
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 10 mg slow intravenous push (bolus) over 5 minutes and then 0.01 mg/kg/min for 55 minutes (Active Comparator): Low dose DMT
  Interventions: Drug: DMT-Low Dose
- 14 mg slow intravenous push (bolus) over 5 minutes and then 0.015 mg/kg/min for 55 minutes. (Active Comparator): Medium Dose DMT
  Interventions: Drug: DMT-Medium Dose
- 0.5 mg over 5 minutes and then 2 mg over and 55 minutes (Active Comparator): THC-Medium Dose
  Interventions: Drug: THC-Medium Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: DMT-Medium Dose; Drug: DMT-Low Dose; Drug: THC-Medium Dose; Drug: THC-Low Dose
- 0.1 mg slow intravenous push (bolus) over 5 minutes and then I mg over 55 minutes (Active Comparator): Low Dose THC
  Interventions: Drug: THC-Low Dose

INTERVENTIONS:
Drug: DMT-Medium Dose — 14 mg slow intravenous push (bolus) over 5 minutes and then 0.015 mg/kg/min for 55 minutes.
  Arms: 14 mg slow intravenous push (bolus) over 5 minutes and then 0.015 mg/kg/min for 55 minutes.; Placebo
Drug: DMT-Low Dose — 10 mg slow intravenous push (bolus) over 5 minutes and then 0.01 mg/kg/min for 55 minutes
  Arms: 10 mg slow intravenous push (bolus) over 5 minutes and then 0.01 mg/kg/min for 55 minutes; Placebo
Drug: THC-Medium Dose — 0.5 mg over 5 minutes and then 2 mg over and 55 minutes
  Arms: 0.5 mg over 5 minutes and then 2 mg over and 55 minutes; Placebo
Drug: THC-Low Dose — 0.1 mg slow intravenous push (bolus) over 5 minutes and then I mg over 55 minutes
  Arms: 0.1 mg slow intravenous push (bolus) over 5 minutes and then I mg over 55 minutes; Placebo

SUMMARY:
The goal of this phase 1 study is to investigate the safety and efficacy of dimethyltryptamine (DMT) in individuals with depression and healthy controls. We hypothesize that administration of DMT will result in decreases in depression, associated symptoms, and neuroplastic changes in depressed subjects. We expect that DMT will induce changes in neuroplasticity as indexed using electroencephalographic (EEG) measures and tasks in both depressed individuals and healthy volunteers, though to different degrees. These neuronal changes may in parallel cause changes in mood measured both in healthy and depressed subjects, which will be captured using appropriate psychometric measures of mood.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age 21 to 65 years;
3. Body mass index between 18-35 kg/m2;
4. English speaking
5. Able to provide informed consent;
6. Willing to refrain from taking any medications not approved by the study physician;
7. Willing to refrain from using street drugs and alcohol the day before, the day of, and the day after each test session;
8. Negative urine drug screen on the morning of each test session (the following drugs will be tested for: cocaine, opioids, benzodiazepines, cannabinoids, stimulants);
9. Willing and able to abstain from smoking throughout each test session;
10. Women who are of child-bearing potential (WOCBP) and sexually active must be willing to practice an effective means of birth control;
11. Willing not to drive to and from the testing session.

Inclusion Criteria for Subjects with MDD:

1. Diagnosed with Major Depressive Disorder (MDD), single or recurrent episode, and currently experiencing a Major Depressive Episode (MDE), of a moderate to severe degree (Score ≥17 on the 21-item clinician-rated HAMD);
2. Unsatisfactory response to at least one adequate antidepressant trial (at least 6 weeks on a therapeutic dose) during the current depressive episode and/or unable to tolerate existing antidepressants, assessed with the Antidepressant Treatment History Form - Short Form (ATHF-SF) and confirmed with the primary mental health provider (see clinician contact form);
3. Engaged in treatment for depression with a clinician and willing to continue treatment for the duration of the study;
4. Those not engaged in treatment t the time of screening will be required to engage in treatment as a condition of study participation.
5. Consent to allow the research team to engage the primary mental health provider.

Exclusion Criteria:

1. Recent clinically significant current risk for suicidal behavior as assessed by chart review, opinion of mental health provider and Columbia Suicide Rating Scale (CSSRS);
2. Recent clinically significant aggressive behavior assessed by chart review, opinion of mental health provider and psychiatric screening;
3. Psychosis:

   1. Current or past history of any psychotic disorder including Schizophrenia, Bipolar I Disorder, Delusional Disorder, Paranoid Personality Disorder, or Schizoaffective Disorder (clinical judgement will be exercised);
   2. History of psychotic symptoms in the current or previous depressive episodes;
4. Currently taking an antidepressant medication (including SSRIs, SNRIs, TCAs, and MAOIs) or other medications (e.g., efavirenz, locanserin) that may alter the effects of 5HT2A agonists. Exceptions are medications used at low doses for sleep. If a subject meets all other study criteria, he/she may consider discontinuation of antidepressant under clinical supervision contingent upon the approval of the patient's clinician. Subjects will need to be off prohibited medications for at least five half-lives of the medication's major metabolites prior to the first test session;
5. Currently taking over the counter products such as 5-hydroxytryptophan and St. John's wort, due to potential interactions with DMT;
6. Cognitive dysfunction that could interfere with study participation;
7. Recent history of meeting criteria for alcohol or substance use disorder (excluding caffeine and nicotine);
8. Alcohol use of ≥7 drinks in females and 14 in males per week (NIAAA guidelines);
9. Any lifetime history of hallucinogen use disorder;
10. Regular (≥once per month) use or misuse of serotonergic hallucinogens including DMT, psilocybin, LSD, and related compounds;
11. History of intolerance to drugs known to significantly alter perception, e.g., DMT, THC ketamine, psilocybin, LSD, Salvinorin A, mescaline, etc.;
12. Hypotension, as defined as a baseline blood pressure < 90/60 mmHg or orthostatic hypotension as defined as a sustained reduction of systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of 10 mm Hg within 3 min of standing or head-up tilt;
13. Pregnancy or currently breast feeding (lactation);
14. Medical conditions deemed by the PI (D'Souza), or his designee, to be unstable including but not limited to uncontrolled hypertension (e.g., >140/90 averaged across four assessments, uncontrolled insulin-dependent diabetes, renal or hepatic failure, seizure disorder, etc.;
15. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation;
16. Any current or past history of any physical condition or abnormal screening laboratory test that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation.
17. First degree relatives with a history of psychosis

IQ < 80 measured by the Weschler Test of Adult Reading (WTAR).Exclusion criteria for depressed subjects:

1. Current primary psychiatric disorder other than MDD;
2. Medically significant condition rendering unsuitability for the study;
3. History of mania;

Exclusion criteria for healthy controls:

1. No current DSM-V psychiatric disorder, excluding nicotine and caffeine use disorder;
2. No lifetime use of psychiatric medication >3 months (proxy for psychiatric disorders).
3. No family history of serious mental illness (e.g., schizophrenia, bipolar disorder)

Inclusion criteria for healthy controls:

1. no current DSM-5 psychiatric disorder, excluding nicotine and caffeine use disorder;
2. no lifetime use of psychiatric medication >3 months (proxy for psychiatric disorders).

Alcohol and street drug use that does not meet criteria for use disorder will be evaluated by the researchers on a case-by-case basis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Physiological indices | Time Frame: -60 and -30 minutes before DMT administration; 0, +5, +10, +15, +20, +30, +45, +60, and +120 minutes after DMT administration]blood pressure and heart rate will be measured before, during, and after the dosing on each test day.
  Pulse oximetry will be measured continuously.
Psychedelic Effects | From start Test Day Time points (Minutes): -60, +30, +120.
  The 30-item revised Mystical Experience Questionnaire (MEQ30) will be used to measure mystical/psychedelic experiences associated with drugs like psilocybin
Psychotomimetic Effects | Test Day Time points (Minutes): -60, +30, +120
  To capture the effects of DMT/THC/placebo on perception, thought, and sensory processing, participants will be measured using the Psychotomimetic States Inventory
Anxiety | Test Day Time points (Minutes): -60, +30, +120
  Will be assessed using a visual analog scale that subjects will be asked to score from 0 (not at all) to 100 (worst ever) to capture anxiety.
Depression | From start of test day (-60), +30, and +120.
  subjects will be asked to score from 0 (not at all) to 100 (worst ever) to capture the depression.
Intensity of the Experience | Test Day Time points (Minutes): +150 - +180
  The Challenging Experience Questionnaire (CEQ) a 26 item likert-scale style survey will be used to provide a phenomenological profile specifically of challenging aspects of experiences with psilocybin
Drug Reinforcing Effects | Test Day Time points (Minutes): +120
  Will be assessed with questions such as:
  * How likely are you to use this drug recreationally? 0 (not at all) ------------------------100 (most of all)
  * How much are you willing to pay for the acute effects that you experienced during the dosing session? $0-------------------$100 Shortly after resolution of effects, participants will be instructed to retroactively rate the highest effects experienced since the last time they were prompted to provide a rating.
Tolerability of Overt Adverse Effects | Test Day Time points (Minutes): -60, +30, +120, 180 (end of test day)
  Tolerability defined by the US FDA as "the degree to which overt adverse effects can be tolerated" by a subject was assessed [60]. At the end of the test day, after all drug effects have worn off, participants will be asked to score 1) the overall experience on a visual analog scale [VAS] (0 = intolerable to 100 = well-tolerated).
Electrophysiological | Resting State EEG: Will be collected the day after each dosing session. [Time Frame: -60 minutes before DMT administration until +180 minutes after DMT administration].

SECONDARY OUTCOMES:
Expectancy Effects | Subjects will be tested for expectancy effects at screening, and before each dosing session.
Adequacy of blinding | Time Frame: 0; immediately after DMT administration, and +180 minutes at the end of the study
  Subjects will be asked to guess their treatment assignment, the degree of certainty of their guess and the reason for their guess both immediately after the psychedelic dosing session(s) and at the end of the study. Either the James' blinding index (BI) or Bang's BI, will be used to measure the adequacy of the blind.
Blood | Blood sample measurements will be repeated approximately 0, 20, 30, and 60 minutes after drug administration
Changes in personality domains (NEO personality inventory) | [Time Frame: -60 minutes before DMT administration; 0, +30, and +60 minutes after DMT administration]
Psychological Flexibility | Time Frame: +180 minutes after DMT administration
  The Acceptance and Action Questionnaire (AAQ) is a one-factor, likert scale assessment of psychological inflexibility

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine,, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No